CLINICAL TRIAL: NCT06119763
Title: Anti-DFS70 Antibodies and it's Relationship With Systemic Lupus Erythematosus Manifestations
Brief Title: AntiDFS70 Lupus Nephritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ashrakat Shabaan Mohamed, resident at rheumatology and rehabilitation department, Sohag University
Other Study IDs: Soh-Med-23-10-011MS
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: systemic lupus erythematosus cases, diagnosed by SLICC criteria with negative levels of AntiDFS antibodies
  Interventions: Diagnostic Test: anti dfs70 antibodies
- group B: systemic lupus erythematosus cases, diagnosed by SLICC criteria with positive levels of AntiDFS antibodies
  Interventions: Diagnostic Test: anti dfs70 antibodies

INTERVENTIONS:
Diagnostic Test: anti dfs70 antibodies — blood sample is taken from SLE cases and is tested for antiDFS70 antibodies titre

SUMMARY:
Systemic lupus erythematous (SLE) is a heterogeneous autoimmune disease that involve many different organs and display a variable clinical course. The prevalence of SLE varies across gender, race/ethnicity, and geographic regions. SLE demonstrates a striking female predominance with a peak incidence of disease during the Reproductive years. In adults, the female to male ratio is 10- 15:1(1)( 2)

Clinical features in individual patients can be quite variable and range from mild joint and skin involvement to severe, life-threatening internal organ disease. Constitutional symptoms, rash, mucosal ulcers, inflammatory polyarthritis, photosensitivity, and serositis are the most common clinical features of the disease. (3) (4) Anti-DFS70 antibodie) and their clinical associations remain an immunological paradox. Unlike other antinuclear antibodies , there is a growing body of evidence that anti-DFS70 antibodies, when present in high titers and in isolation (without accompanying other antibodies), are useful to aid in the exclusion of antinuclear antibodies associated rheumatic diseases. (8)

Anti-DFS70 antibodies were not associated with lupus nephritis development in Systemic lupus erythematosus patients but were associated with anti-dsDNA antibodies , proliferative lupus nephritis, and renal activity index . This suggests their potential to serve as a non-histological biomarker for lupus nephritis subclass and activity status. (8)

ELIGIBILITY:
Inclusion Criteria:

1. Patients who fulfill the 2019 American College of Rheumatology/European League against Rheumatism classification criteria of Systemic Lupus Erythematous . (9)
2. Patients who is able to give informed consent to join the study.

   •

   Exclusion Criteria:

   -

   - Any patient with any collagen disease other than systemic lupus erythematous

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Patients who fulfill the 2019 American College of Rheumatology/European League against Rheumatism classification criteria of Systemic Lupus Erythematous . (9)
  2. Patients who is able to give informed consent to join the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
antiDFS70 antibodies titre | 1 year
  serve as a non-histological biomarker for lupus nephritis subclass and activity status.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pons-Estel GJ, Alarcon GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010 Feb;39(4):257-68. doi: 10.1016/j.semarthrit.2008.10.007. Epub 2009 Jan 10. PMID 19136143
- [Background] Lim SS, Bayakly AR, Helmick CG, Gordon C, Easley KA, Drenkard C. The incidence and prevalence of systemic lupus erythematosus, 2002-2004: The Georgia Lupus Registry. Arthritis Rheumatol. 2014 Feb;66(2):357-68. doi: 10.1002/art.38239. PMID 24504808
- [Background] DUBOIS EL, TUFFANELLI DL. CLINICAL MANIFESTATIONS OF SYSTEMIC LUPUS ERYTHEMATOSUS. COMPUTER ANALYSIS OF 520 CASES. JAMA. 1964 Oct 12;190:104-11. doi: 10.1001/jama.1964.03070150014003. No abstract available. PMID 14184513
- [Background] Hahn BH, McMahon MA, Wilkinson A, Wallace WD, Daikh DI, Fitzgerald JD, Karpouzas GA, Merrill JT, Wallace DJ, Yazdany J, Ramsey-Goldman R, Singh K, Khalighi M, Choi SI, Gogia M, Kafaja S, Kamgar M, Lau C, Martin WJ, Parikh S, Peng J, Rastogi A, Chen W, Grossman JM; American College of Rheumatology. American College of Rheumatology guidelines for screening, treatment, and management of lupus nephritis. Arthritis Care Res (Hoboken). 2012 Jun;64(6):797-808. doi: 10.1002/acr.21664. No abstract available. PMID 22556106